CLINICAL TRIAL: NCT00569777
Title: A Multi-Center, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Study Evaluating the Safety of a Novel Contact Lens Used Daily in Healthy, Normal Volunteers
Brief Title: Safety Study of a Contact Lens With Ketotifen in Healthy, Normal Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 07-003-002
Record Dates: First submitted 2007-11-27; First posted 2007-12-07 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- K-lens (Experimental): etafilcon A contact lens with ketotifen.
  Interventions: Device: K-Lens (generic name not established) and Ketotifen
- Placebo (Placebo Comparator): etafilcon A contact lens without ketotifen
  Interventions: Device: Placebo Lens

INTERVENTIONS:
Device: K-Lens (generic name not established) and Ketotifen — combination drug-device product: contact lens (device) and anti-allergy drug
  Arms: K-lens
Device: Placebo Lens — contact lens without drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of a novel contact lens in healthy normal volunteers

ELIGIBILITY:
Inclusion Criteria:

* healthy normal, soft contact lens wearing volunteers
* normal ocular health
* contact lens correction from +6.00 to -12.00D in each eye and astigmatism of -1.00D or less in each eye

Exclusion Criteria:

* active ocular infection
* history of ocular surgery
* use of topical ophthalmic preparations (including rewetting drops)
* pregnancy or lactation

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pall, OD, MS, FAAO, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (3):
- United States (3):
  - Gardena, California
  - North Andover, Massachusetts
  - Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | K-lens | Placebo
Started | 206 | 104
Completed | 196 | 101
Not Completed | 10 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — scheduled eye surgery | 0 | 1
Not completed — did not meet exclusion criteria | 1 | 2
Not completed — pregnant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | K-lens | Placebo | Total
Number analyzed (Participants) | 206 | 104 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11.62) | 30 (10.75) | 31 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 80 | 224
  Male | 62 | 24 | 86
Region of Enrollment [Number; unit: participants]
  United States | 206 | 104 | 310

OUTCOME MEASURES:

1. Primary Outcome: Lid and Lid Margin Erythema, Change From Baseline
Description: Assessment of lid redness using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.053) | 0 (0.129)

2. Primary Outcome: Lid and Lid Margin Swelling, Change From Baseline
Description: Assessment of lid swelling using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 104
Number analyzed (eyes) | 362 | 208
Units on a scale | 0 (0) | 0 (0)

3. Primary Outcome: Conjunctival Redness, Change From Baseline
Description: Assessment of redness of conjunctiva using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.632) | -0.1 (0.522)

4. Primary Outcome: Conjunctival Chemosis, Change From Baseline
Description: Assessment of swelling of the conjunctiva using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 177
Units on a scale | 0 (0.105) | 0 (0.166)

5. Primary Outcome: Corneal Edema, Change From Baseline
Description: Assessment of corneal swelling using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0) | 0 (0)

6. Primary Outcome: Corneal Erosion, Change From Baseline
Description: Assessment of corneal erosion using the following scale: 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0) | 0 (0.106)

7. Primary Outcome: Corneal Endothelial, Change From Baseline
Description: Assessment of the posterior cornea using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Analysis includes subjects that completed the 12 week visit per protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0) | 0 (0)

8. Primary Outcome: Lens Pathology, Change From Baseline
Description: Assessment of the clarity of the intraocular lens using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.181) | -0.1 (0.254)

9. Primary Outcome: Flare in Anterior Chamber, Change From Baseline
Description: Assessment of visible protein in the anterior chamber using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0) | 0 (0)

10. Primary Outcome: Cells in Anterior Chamber, Change From Baseline
Description: Assessment of visible cells in the anterior chamber using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0) | 0 (0)

11. Primary Outcome: Corneal Staining - Nasal, Change From Baseline
Description: Assessment of changes to the surface of cornea, the region towards the nose, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | -0.1 (0.28) | 0 (0.35)

12. Primary Outcome: Corneal Staining - Temporal, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the region towards the outer edge of the face, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.271) | 0 (0.256)

13. Primary Outcome: Corneal Staining - Inferior, Change From Baseline
Description: Assessment of changes to the surface of the cornea, the bottom region, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.515) | 0 (0.53)

14. Primary Outcome: Corneal Staining - Superior, Change From Baseline
Description: Assessment of changes to the surface of the cornea, upper region, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.229) | 0 (0.149)

15. Primary Outcome: Corneal Staining - Central, Change From Baseline
Description: Assessment of changes to the surface of the cornea, central region, as evaluated by the degree of staining with sodium fluorescein solution, using the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Units on a scale | 0 (0.234) | 0 (0.212)

16. Primary Outcome: Intraocular Pressure, Change From Baseline
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: mm of mercury
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
mm of mercury | -0.3 (2.7) | -0.4 (2.707)

17. Primary Outcome: Dilated Ophthalmoscopy - Fundus, Change From Baseline
Description: Assessment of changes in abnormalities on the back part of the eye, using the scale: 0=none, 0.5=trace, 1=mild, 2=moderate, 3=severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis. K-lens: missing data for 2 subjects/4 eyes.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 179 | 89
Number analyzed (eyes) | 358 | 178
Units on a scale | -0.1 (0.371) | 0 (0.235)

18. Primary Outcome: Dilated Ophthalmoscopy - Vitreous, Change From Baseline
Description: Assessment of changes in the vitreous (gel-like fluid of the eye), using the scale: 0=none, 0.5=trace, 1=mild, 2=moderate, 3=severe.
Time Frame: baseline and 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis. K-lens: missing data for 2 subjects / 4 eyes.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 179 | 89
Number analyzed (eyes) | 358 | 178
Units on a scale | 0 (0.149) | 0 (0.149)

19. Primary Outcome: Visual Acuity Assessment
Description: Visual acuity was assessed by the investigator using a Snellen visual acuity chart. This outcome counts the number of eyes that had vision of 20/40 or better at the 12 week visit.
Time Frame: at 12 weeks
Population: Subjects that completed the study per protocol were included in this analysis.
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | K-lens | Placebo
Number analyzed (Participants) | 181 | 89
Number analyzed (eyes) | 362 | 178
Eyes | 362 | 178

ADVERSE EVENTS:
Arm/Group | K-lens | Placebo
Serious Adverse Events (participants affected / at risk) | 2/206 | 0/104
Other Adverse Events (participants affected / at risk) | 11/206 | 4/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | K-lens (N=206) | Placebo (N=104)
nasal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — nasal fracture resulting from an accident, unrelated to test article
abdominal discomfort requiring hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) — unrelated to test article
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-lens (N=206) | Placebo (N=104)
nasopharyngitis (Infections and infestations) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish or publicly present the data and or results of the study without prior approval from Vistakon.